CLINICAL TRIAL: NCT02853461
Title: Biofilm Investigation on Ceramic, Metal and Polyethylene Bearing Components From Explanted Hip Joint Prosthesis
Brief Title: Biofilm Investigation on Bearing Components of Explanted Hip Joint Prosthesis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Ceram Tec GmbH (Unknown); Pro-Implant Foundation (Other)
Responsible Party: Principal Investigator, Andrej Trampuz, MD, Charite University, Berlin, Germany
Other Study IDs: Endo 015/15
Record Dates: First submitted 2016-07-20; First posted 2016-08-03 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Sonication; Total Hip Replacement; Biofilm
Keywords: biofilm; periprosthetic joint infection; hip; endoprothesis; ceramic; bearing components; sonication; low grade infection; joint aspiration
MeSH Terms: interventions — Sonication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Sonication — Ultrasound bath (40 kHz, 1 W/cm2, 1 min) of bearing components of the prosthesis in sterile conditions.
Other: Microbiological analysis — Plating the sonicates on agar plates.

SUMMARY:
In this study the investigators sonicate the bearing components of the explanted hip prosthesis which allows highly sensitive detection of in vivo biofilms (qualitatively and quantitatively). The hip prosthesis bearing components are composed from different material. The purpose of this study is to analyse the resistance against biofilm adhesion of ceramic, metal and polyethylene prosthesis components through microbiologic analysis of sonicates.

DETAILED DESCRIPTION:
The main reasons for hip prosthesis failure are aseptic loosening and periprosthetic joint infection (PJI). The real frequency of PJI is probably largely underestimated because of non-standardized definition criteria, diagnostic procedure, treatment algorithm and other confounders. Therefore, data from joint registries are not reflecting the frequency of PJI and can be misleading; particularly low-grade PJI can be frequently misdiagnosed as aseptic failure.

Microbiological analysis of sonicate has in comparison with joint aspirate significantly higher sensitivity and specificity, which allows better detection of low grade infection. With aspiration only free-floating, high metabolically active, planktonic form of bacteria could be collected. Contrarily, the less metabolically active bacteria are hidden under the biofilm can remain undetected.

Sonication of prosthetic material mechanically dislodge the biofilm from surface and expose the sessile bacteria for the microbiological analysis.

All foreign materials provoke biofilm formation however, different materials showed different resistance for biofilm adhesion.

In this study patients with PJI are undergoing standard one- or two- stage revision procedure of the hip. The removed bearing components will be sonicated and sent in microbiological analysis. The ceramic, metal and polyethylene prosthesis components will undergo qualitative and quantitative microbiological analysis. The materials will be compared regarding to the presence of biofilm formation.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be aged 18 or more.
* Subject must be scheduled to undergo an explanation of the hip endoprosthesis during the 1- or 2- stage revision procedure because of the septic or mechanical indication.
* Subject must personally sign and date the informed consent document indicating that the subject has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Patient not scheduled for the index Operation procedure with removal of hip endoprosthesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥18 y, undergoing hip prosthesis explantation for infection or mechanical (aseptic) reason.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Qualitative analysis of sonication fluid after sonication of explanted bearing components of the hip endoprosthesis during a revision surgery | Prospective: patient recruitment up to 2 years
  Qualitative Analysis, i.e. frequency of positive sonication fluid cultures (No. positive/No. all cultures) deriving from 3 different biomaterials (namely: Ceramic, Cobalt-chrome-metal, and Polyethylene), the number of variables which will be evaluated following: bearing component and its material (Ceramic, Cobalt-chrome-metal, and Polyethylene).
  All three material types will be compared between each other regard to microbiology analysis of sonication fluid of bearing components.
Quantitative Analysis e.g. No. of microorganisms in sonication fluid (CFU/ml) deriving from 3 different biomaterials (namely: Ceramic, Cobalt-chrome-metal, and Polyethylene). | Prospective: patient recruitment up to 2 years

SECONDARY OUTCOMES:
Amount of patients with septic loosening of hip joint | Prospective: patient recruitment up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Trampuz, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Achermann Y, Vogt M, Leunig M, Wust J, Trampuz A. Improved diagnosis of periprosthetic joint infection by multiplex PCR of sonication fluid from removed implants. J Clin Microbiol. 2010 Apr;48(4):1208-14. doi: 10.1128/JCM.00006-10. Epub 2010 Feb 17. PMID 20164283
- [Background] Banche G, Allizond V, Bracco P, Bistolfi A, Boffano M, Cimino A, Brach del Prever EM, Cuffini AM. Interplay between surface properties of standard, vitamin E blended and oxidised ultra high molecular weight polyethylene used in total joint replacement and adhesion of Staphylococcus aureus and Escherichia coli. Bone Joint J. 2014 Apr;96-B(4):497-501. doi: 10.1302/0301-620X.96B4.32895. PMID 24692617
- [Background] Gomez-Barrena E, Esteban J, Medel F, Molina-Manso D, Ortiz-Perez A, Cordero-Ampuero J, Puertolas JA. Bacterial adherence to separated modular components in joint prosthesis: a clinical study. J Orthop Res. 2012 Oct;30(10):1634-9. doi: 10.1002/jor.22114. Epub 2012 Mar 30. PMID 22467526